CLINICAL TRIAL: NCT06397885
Title: Prospective on Market Patient-reported Outcomes for Milli
Acronym: POMPOM
Status: Active, not recruiting | Type: Observational
Sponsor: Materna Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CP0004
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Vaginismus; Dyspareunia
Keywords: painful sex; dilation
MeSH Terms: conditions — Vaginismus; Dyspareunia; Dilatation, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Milli Vaginal Dilator — Patient-controlled vaginal dilator that provides therapy through distention of the vaginal tissue under electromechanical expansion

SUMMARY:
To assess the effectiveness of the Milli device in achieving vaginal intercourse

DETAILED DESCRIPTION:
The Milli Vaginal Dilator is a patient-controlled vaginal dilator that provides therapy through distention of the vaginal tissue under electromechanical expansion.

This study is intended to provide data in support of the Milli Vaginal Dilator as a commercially available, over-the-counter medical device.

The Milli has been granted marketing authorization by the FDA under premarket notification K220035 for the following Indications for Use statement:

The Milli Vaginal Dilator is a tool indicated for controlled dilation of the vagina. It can be used for dilation for an examination (by your doctor), in preparation for a surgical procedure, or to help relieve the symptoms of vaginismus (condition that involves tightening of the vaginal muscles) and related painful sex.

.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female at birth aged ≥18 years of age
* Subject is able to read and understand the approved, informed consent form (ICF)
* Subject meets vaginismus and related painful sex/GPPPD criteria as defined in the DSM-5, as confirmed by having one or more of the following for greater than 6 months:
* Pelvic pain
* Vaginal pain
* Pain with vaginal intercourse
* Pain with vaginal penetration
* Fear or anxiety about vaginal or pelvic pain with vaginal penetration
* The inability to achieve vaginal penetration
* Subject currently has a sexual partner with a functional penis
* Subject is currently seeking vaginal penetration to achieve sexual intercourse
* Subject is currently unable to tolerate vaginal penetration to achieve sexual intercourse (Score of ≤1 on PEQ Question #1)
* Subject purchased Milli vaginal dilator
* Subject is not contraindicated for Milli vaginal dilator use
* Subject is able and willing to comply with study protocol

Exclusion Criteria:

* Subject has previously participated in any studies by the company in the past 12 months or has used Milli prior to enrollment
* Subject is pregnant
* Subject has an active pelvic infection (vagina or vulva)
* Subject has open wounds in the tissue inside or surrounding the vagina
* Subject has an untreated major mental health disorder (e.g., affective disorder, psychosis, PTSD)
* Subject has prior history of gender-confirming surgery, vaginal reconstruction surgery, pelvic radiation, and/or vaginal procedures that result in extensive scarring (with the exception of hysterectomy procedures)
* Subject or subject's partner experiences other conditions preventing intercourse (e.g., erectile dysfunction, lack of libido)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects eligible if female at birth, aged ≥18 years
Study Population: The study population shall include subjects seeking relief for the symptoms of vaginismus and/or associated dyspareunia (painful sex).
  The Milli Vaginal Dilator is cleared for use as an Over-The-Counter device (K220035). As such, the study population shall be comprised of all adult subjects who provide (≥18 years of age) Informed Consent.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Penetration Efficiency Questionnaire | 6 months
  Ability to achieve full vaginal penetration with the penis of the partner (intercourse) as measured by the Penetration Efficiency Questionnaire (Score of ≥2 on PEQ Question #1) at six months

SECONDARY OUTCOMES:
Penetration Efficiency Questionnaire | 3 months
  Ability to achieve full vaginal penetration with the penis of the partner (intercourse) as
Penetration Efficiency Questionnaire | 3 months, 6 months
  Improvement in ability to achieve vaginal penetration (intercourse and non-intercourse) as measured by a change in baseline in the overall score on the Penetration Efficiency Questionnaire at 3 and 6 months.
Female Sexual Function Index (FSFI) | 3 months, 6 months
  Improvement in self-reported sexual function as reported on a change in baseline in the Female Sexual Function Index (FSFI) total score at 3 and 6 months.
Numerical Rating Scale | 3 months, 6 months
  Improvement in self-reported pain intensity with intercourse as reported as a change in baseline on a numeric rating scale (NRS) (0= no pain, 10 = worst pain imaginable) at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl Kingsberg, Ph.D, Principal Investigator — Materna Clinic
Locations (1):
- Materna Clinic, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No